CLINICAL TRIAL: NCT04400812
Title: Attitude and Perception of General Population in Sharkia Governerate Towards COVID-19 Pandemic
Brief Title: Attitude and Perception Towards COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Waheed Shouman, professor of chest diseases, Zagazig University
Other Study IDs: ZU#IRB#6138-17-5-2020
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — Arabic questionnaire focused on knowledge, perception and attitude

SUMMARY:
Assess response and attitude of general population living in Sharkia Governerate, Egypt as regard COVID-19 pandemic through arabic questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* General population within age range (16-70) and both sexes living in Sharkia Governerate, Egypt and accept to participate

Exclusion Criteria:

* below 16 or above 70 years
* refuse to participate
* duplicate answers
* incomplete answers

Ages: 16 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: General population within age range (16-70) and both sexes living in Sharkia Governerate, Egypt and accept to participate
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-05-19 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Knowledge about COVID-19 by questionnaire | 30 days after enrollment
Perception about COVID-19 by questionnaire | 30 days after enrollment
Attitude towards COVID-19 by questionnaire | 30 days after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University, Zagazig, Sharqia Province, Egypt